CLINICAL TRIAL: NCT00390663
Title: A Prospective Randomised Controlled Trial of Management of Recurrent Nosebleeds in Children: Antiseptic Cream Alone v's Antiseptic Cream With Nasal Cautery
Brief Title: A Prospective Randomised Controlled Trial of Management of Recurrent Nosebleeds in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow Yorkhill Division (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 05/EN/03
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2006-10

CONDITIONS: Epistaxis
Keywords: Paediatric; Epistaxis; Nose bleed; Naseptin
MeSH Terms: conditions — Epistaxis

INTERVENTIONS:
Procedure: Nasal Cautery

SUMMARY:
To determine whether the selective application of a combined treatment regimen of silver nitrate cautery and 4 weeks of Naseptin cream is superior to naseptin treatment alone in the management of recurrent paediatric epistaxis.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 - 14
* History of repeated epistaxis with at least 1 episode in the previous 4 weeks prior to attending the ENT clinic.
* Presence of prominent vessels on the anterior nasal septum on the side that reportedly bleeds (or on at least one side if bleeding is reported to be bilateral)

Exclusion Criteria:

* No prominent vessels on examination (these children will be randomised but will be prescribed Naseptin alone and followed up in the same way as the children in the trial, for completeness of data)
* Known bleeding disorders.
* Allergy to peanuts, neomycin or chlorhexidine
* Other causes of nose bleeding eg tumour.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Haytham Kubba, MBBS(Hons) MPhil FRCS FRCSEd, Principal Investigator — Royal Hospital for Sick Children
Locations (1):
- Royal Hospital for Sick Children, Glasgow, Strathclyde, United Kingdom